CLINICAL TRIAL: NCT04159220
Title: Randomized Controlled Trial to Evaluate an Optimization Procedure of Alveolar Recruitment During Transport Performed by Nurse Anesthetists in Intensive Care
Brief Title: Trial to Evaluate an Optimization Procedure of Alveolar Recruitment During Transport Performed by Nurse Anesthetists in Intensive Care
Acronym: ESCORTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RECHMPL19_0070
Record Dates: First submitted 2019-11-06; First posted 2019-11-12 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Respiratory Complication

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The transport will be released without a clamping of endotracheal tube before each disconnection from ventilator.
- Clamping group (Experimental): The transport will be released with a clamping of endotracheal tube before each disconnection from ventilator.
  Interventions: Procedure: Clamping of the ventilator endotracheal tube

INTERVENTIONS:
Procedure: Clamping of the ventilator endotracheal tube — The transport will be released in accordance with SFAR SRLF guideline. Before each disconnection from ventilator endotracheal tube will be clamped.
  Arms: Clamping group

SUMMARY:
Intra hospital transport of ICU patients is still at high risk of respiratory complications.We propose to determine if endotracheal tube clamping prior to disconnect ventilator allows to avoid oxygenation decrease.

DETAILED DESCRIPTION:
Changing respiratory support and multiples endotracheal tube disconnections may induce a loss of PEEP and finally lead to alveolar derecruitment. This study is an evaluation of a care procedure to limit the incidence of alveolar derecruitment in ventilated intubated ICU patients during transport for CT scan.

Intra hospital transport of ICU patients are performed by anesthesiologist nurses, the physician entrusts them this activity.

This is a randomized controlled study, the procedure is to clamp endotracheal tube before each disconnection from ventilator.

ELIGIBILITY:
Inclusion Criteria:

* intensive care patient
* intubated, sedated, controlled assisted ventilation
* Intra hospital transport for CT scan
* arterial catheter
* the patient or his trusted person consent to the study

Exclusion Criteria:

* Patient Covid tests positive or Covid test results not received
* extubated, unsedated,
* reinforced tube
* tracheotomy
* pregnancy
* guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Measure of the pa02/Fi02 | 1 hour after the end of the transport
  Evaluate the effectiveness of a procedure to avoid alveolar delisting, measured by the absence of a decrease in the PaO2/FiO2 ratio (before transport and 1 hour after return to bed) during an HIT performed by a nurse anaesthetist/caregiver team, of intubated and ventilated resuscitation patients in a controlled assisted volume.

SECONDARY OUTCOMES:
Assessment of the pa02 | 1 hour after the end of the HIT
  Evaluate the impact of the procedure on the absence of PaO2 reduction (before transport and 1 hour after return to bed)
Assessment of the pa02 | immediately after the end of the HIT
  Evaluate the effectiveness of the procedure on Pa02 immediately after reconnection to the heavy resuscitation ventilator
Assessment of the pa02 | 6 hours after the end of of the HIT
  Evaluate the effectiveness of the procedure on Pa02 immediately after reconnection to the heavy resuscitation ventilator
length of stay | up to 28 days
  Evaluate the impact of the intervention on the length of ICU stay
duration of invasive ventilation | up to 28 days
  Evaluate the impact of the intervention on the invasive ventilation
occurrence of adverse events during the HIT | immediately after the end of the HIT
  occurrence of adverse events related to the clamping

CONTACTS AND LOCATIONS:
Locations (1):
- Departement d'anesthésie et réanimation Gui de Chauliac (DAR C), Montpellier, France

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: 12 months after the main publication
Access Criteria: Data are provided to qualified investigators free of charge. Required documents to request data include a summary of the research plan, request form, and IRB review. Dataset will be shared after careful examination by the study board of investigators.